CLINICAL TRIAL: NCT06532682
Title: Efficacy and Mechanism of Dapagliflozin Combined With Insulin in the Treatment of Early Diabetic Nephropathy in Patients With Type 1 Diabetes
Brief Title: Efficacy of Dapagliflozin in Early Diabetic Nephropathy in Type 1 Diabetes
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-SR-929
Record Dates: First submitted 2024-07-23; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Diabetic Kidney Disease; Type 1 Diabetes
MeSH Terms: conditions — Diabetic Nephropathies; Diabetes Mellitus, Type 1 | interventions — dapagliflozin; Angiotensin-Converting Enzyme Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Drug: Dapagliflozin 10 MG + ACE inhibitor (Experimental): Using ACE inhibitors/ARBs as standard treatment, dapagliflozin is administered at a dose of 10 mg once daily, without food restrictions, for a total treatment duration of 24 weeks.
  Interventions: Drug: dapagliflozin; Drug: ACE inhibitor
- Drug: Dapagliflozin 5 MG + ACE inhibitor (Experimental): Using ACE inhibitors/ARBs as standard treatment, dapagliflozin is administered at a dose of 5 mg once daily, without food restrictions, for a total treatment duration of 24 weeks.
  Interventions: Drug: dapagliflozin; Drug: ACE inhibitor
- Drug: ACE inhibitor (Active Comparator): Using ACE inhibitors/ARBs as standard treatment for a total treatment duration of 24 weeks.
  Interventions: Drug: ACE inhibitor

INTERVENTIONS:
Drug: dapagliflozin — dapagliflozin 5 MG/10 MG once daily
  Other Names: Farxiga
  Arms: Drug: Dapagliflozin 10 MG + ACE inhibitor; Drug: Dapagliflozin 5 MG + ACE inhibitor
Drug: ACE inhibitor — ACE inhibitor

SUMMARY:
Diabetic kidney disease (DKD) is a leading cause of chronic and end-stage kidney disease, affecting 25-40% of type 1 diabetes (T1D) patients and 5-40% of type 2 diabetes (T2D) patients. Despite standard treatments like ACE inhibitors and ARBs, many patients continue to develop DKD, indicating a need for better kidney protection. This study aims to evaluate the efficacy and safety of dapagliflozin combined with insulin in early DKD patients with T1DM, using ACEi/ARB as standard treatment, to provide new insights into kidney protection and support precision medicine goals.

DETAILED DESCRIPTION:
This is an open-label, randomized, parallel-group study to evaluate the effects of dapagliflozin on urinary albumin/creatinine ratio (UACR) in participants with early diabetic nephropathy and type 1 diabetes mellitus (T1DM). The primary objective is to assess the changes in UACR and estimated glomerular filtration rate (eGFR) before and after dapagliflozin treatment in these patients. Secondary objectives include observing blood glucose control, weight improvement, and safety evaluation after dapagliflozin treatment.

The study comprises three groups: dapagliflozin 10 mg, dapagliflozin 5 mg, and a standard treatment control, with a 1:1:1 allocation ratio. Participants meeting the inclusion criteria and not meeting any exclusion criteria will enter a 4-8 week lead-in period, during which they will receive the maximum tolerable dose of ACEI/ARB medications, maintain this treatment for at least 4 weeks, and optimize blood glucose control under the guidance of medical professionals while wearing continuous glucose monitoring devices. Starting from baseline, participants will receive either dapagliflozin 5 mg or 10 mg once daily for 24 weeks, while the control group will continue on the maximum tolerable dose of ACEI/ARB medications. Continuous glucose monitoring and regular ketone monitoring will be performed to prevent diabetic ketoacidosis. Follow-up visits will occur approximately 30 days after the last dose of study medication or upon study completion.

The primary efficacy indicators are the mean changes in UACR and eGFR from baseline to week 24. Secondary efficacy indicators include changes in 24-hour urine biochemistry, HbA1c, body weight, continuous glucose monitoring indices, and total daily insulin dose. Safety evaluation indicators include adverse events, serious adverse events, diabetic ketoacidosis, severe hypoglycemia, and urinary or genital infections.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years;
* Diagnosed with type 1 diabetes mellitus with a disease duration of more than 5 years;
* Glycated hemoglobin (HbA1c) ≤ 7.5% at screening;
* Diagnosed with diabetic nephropathy;
* UACR between 30 and 300 and eGFR ≥ 60 ml/min/1.73 m².

Exclusion Criteria:

* Other types of diabetes;
* Use of any antidiabetic medications (excluding insulin) within 1 month prior to screening;
* History of diabetic ketoacidosis within 3 months prior to screening, or a diagnosed episode of diabetic ketoacidosis within the past 1 month;
* History of poor blood glucose control requiring hospitalization (due to hyperglycemia or hypoglycemia) within 1 month prior to screening;
* Frequent severe hypoglycemia or unconscious hypoglycemia (more than once requiring medical intervention or emergency care) within 1 month prior to screening;
* Use of SGLT2 inhibitors or other renal protective medications within 6 months prior to screening;
* Women who are planning to become pregnant, pregnant, or breastfeeding;
* Cardiovascular disease (within 6 months prior to screening);
* Unstable/rapidly progressing renal disease (within 6 months prior to screening), or renal artery stenosis;
* Major liver disease or malignant tumors (within 5 years prior to screening).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Urinary albumin-to-creatinine ratio | From baseline to 24 weeks
  Average change from baseline to 24 weeks after treatment
estimated Glomerular Filtration Rate | From baseline to 24 weeks
  Average change from baseline to 24 weeks after treatment

SECONDARY OUTCOMES:
24-hour urine biochemical quantification | From baseline to 24 weeks
  Average change from baseline to 24 weeks after treatment
HbA1c | From baseline to 24 weeks
  Change from baseline to 24 weeks after treatment
Weight | From baseline to 24 weeks
  Change from baseline to 24 weeks after treatment
Time in Range | From baseline to 24 weeks
  Evaluate blood glucose control through continuous glucose monitoring
Daily insulin dose | From baseline to 24 weeks
  Change from baseline to 24 weeks after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Mei Zhang, Principal Investigator — Nanjing Medical University First Affiliated Hospital
Locations (1):
- Nanjing Medical University First Affiliated Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No